CLINICAL TRIAL: NCT03375554
Title: The Effect of Esophageal Temperature Probe Insertion on Tracheal Cuff Pressure
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Collaborators: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jung-Man Lee, Clinical assistant professor, Seoul National University Hospital
Other Study IDs: 16-2017-78
Record Dates: First submitted 2017-12-13; First posted 2017-12-18 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-08

CONDITIONS: Intubation Complication
Keywords: esophageal steothoscope, tracheal intubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective observational study is to investigate the effect on esophageal stethoscope insertion on tracheal cuff pressure during general anesthesia.

DETAILED DESCRIPTION:
It is well known that cuff pressure of tracheal tube should not be over 30 cmH2O. Therefore, anesthesiologists usually pay attention to maintain adequate cuff pressure, especially just after completion of tracheal intubation. Recently, esophageal stethoscope is widely used for exact monitoring of patient's body temperature. However, inserting of foreign body in esophagus could affect on the cuff pressure.

The goal of this prospective observational study is to investigate the effect on esophageal stethoscope insertion on tracheal cuff pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patient receiving general anesthesia for elective surgery

Exclusion Criteria:

* who doesn't agree to enroll
* who has any clinical disease or history of surgery in esophagus
* who has aspiration tendency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient receiving general anesthesia for elective surgery
Sampling Method: Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-06-05 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Change of cuff pressure | intraoperative
  Change of cuff pressure by inserting of esophageal stethoscope, compared with before insertion of it

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Man Lee, M.D.,PhD, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Seoul Metropolitan Government Seoul National University Boramae Medical Center, Seoul, South Korea